CLINICAL TRIAL: NCT01338402
Title: Evaluation of the Performance of AIR OPTIX® COLORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: P-368-C-108; P/363/10/C (Other: University of Waterloo)
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AIR OPTIX® AQUA (Other): Lotrafilcon B contact lenses worn in both eyes on a daily wear basis for one week in Phase 1.
  Interventions: Device: Lotrafilcon B contact lens
- AIR OPTIX® COLORS (Experimental): Lotrafilcon B contact lens with color randomly assigned to one eye, with phemfilcon A contact lens with color in the fellow eye for contralateral wear. Both products worn on a daily wear basis for 4 weeks in Phase 2. A replacement phemfilcon A lens was dispensed at the Week 2 visit.
  Interventions: Device: Lotrafilcon B contact lens with color
- FRESHLOOK® COLORBLENDS (Active Comparator): Phemfilcon A contact lens with color randomly assigned to one eye, with lotrafilcon B contact lens with color in the fellow eye for contralateral wear. Both products worn on a daily wear basis for 4 weeks in Phase 2. A replacement phemfilcon A lens was dispensed at the Week 2 visit.
  Interventions: Device: Phemfilcon A contact lens with color

INTERVENTIONS:
Device: Lotrafilcon B contact lens — Silicone hydrogel contact lens
  Other Names: AIR OPTIX® AQUA
  Arms: AIR OPTIX® AQUA
Device: Lotrafilcon B contact lens with color — Silicone hydrogel contact lens with color
  Other Names: AIR OPTIX® COLORS
  Arms: AIR OPTIX® COLORS
Device: Phemfilcon A contact lens with color — Hydrogel contact lens with color
  Other Names: FRESHLOOK® COLORBLENDS
  Arms: FRESHLOOK® COLORBLENDS

SUMMARY:
The purpose of this study was to assess the ocular response to and performance of the cosmetically printed silicone hydrogel contact lens AIR OPTIX® COLORS compared to FRESHLOOK® COLORBLENDS.

DETAILED DESCRIPTION:
The study was conducted in two phases. Phase 1 was an adaptation phase where participants wore AIR OPTIX® AQUA contact lenses bilaterally (same product in both eyes) on a daily wear basis for 1 week. In Phase 2, participants wore AIR OPTIX® COLORS and FRESHLOOK® COLORBLENDS contact lenses contralaterally (different product in each eye) on a daily wear basis for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Full legal capacity to volunteer;
* Read and sign information and consent letter;
* Willing and able to follow instructions and maintain the appointment schedule;
* Ocular examination in the last two years;
* Currently wears soft contact lenses on a daily wear basis;
* Contact lens prescription between -1.50 diopters and -5.00 diopters;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular disease;
* Any systemic condition that may affect a study outcome variable;
* Any systemic or topical medications that may affect ocular health;
* Known sensitivity to the diagnostic pharmaceuticals used in the study;
* Unable to achieve an acceptable fit with the study lenses;
* Anisometropia >1.00 diopter or astigmatism >0.75 diopter;
* Use of lubricating/rewetting eye drops.
* Other protocol-defined exclusion criteria may apply.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | Phase 2: Up to Week 4
Corneal Staining | Phase 2: Up to Week 4
Conjunctival Staining | Phase 2: Up to Week 4
Surface Regularity Index (SRI) | Up to Phase 2, Week 4
Surface Asymmetry Index (SAI) | Up to Phase 2, Week 4
Subjective ratings | Phase 2: Up to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, MOptom, FAAO, Principal Investigator — University of Waterloo Centre for Contact Lens Research; Lyndon Jones, PhD, FCOptom, FAAO, Principal Investigator — University of Waterloo Centre for Contact Lens Research
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada